CLINICAL TRIAL: NCT03215082
Title: Seeing-Moving-Playing: Early Rehabilitation Utilizing Visual and Vestibular Technology Following Traumatic Brain Injury
Acronym: SiMPlyRehab
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Isabelle Gagnon, Clinical Scientist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-3373
Record Dates: First submitted 2017-07-09; First posted 2017-07-12 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Mild Traumatic Brain Injury; Concussion
MeSH Terms: conditions — Brain Concussion | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The intervention will be an individualized impairment-based program based on a pre-determined sequence. A minimal intervention for all participants randomized to the intervention group at all sites will include general oculomotor and gaze stabilization retraining as tolerated. Intervention activities will be recorded and described in detail in a treatment log.
  Interventions: Other: Vestibular-Visual Intervention
- Control (Active Comparator): Standard care for mild TBI consists mainly of general education, energy conservation, academic adaptations, and restricting children and adolescents from participation in vigorous physical activities as well as complex cognitive activities until complete symptom resolution. It is the usual approach promoted by various associations and consensus groups. In addition, in all participating centers, children and teens requiring musculoskeletal approaches to address neck pain/dysfunction will receive it as indicated, based on the clinical judgment of the local team. Participants with moderate and severe TBI will also receive rehabilitation activities as planned in their respective centers. The standard care intervention will be recorded and described in detail in a treatment log.
  Interventions: Behavioral: standard care

INTERVENTIONS:
Other: Vestibular-Visual Intervention — vestibular-visual exercises
  Arms: Experimental
Behavioral: standard care — standard care
  Arms: Control

SUMMARY:
The aim of this research program is to 1) Evaluate potential problems with vision, inner ear-eye reflexes and deficits of processing eye information that occur following TBI; and 2) Evaluate treatment programs for individuals with eye and inner ear problems that persist for greater than 10 days following injury.

This study will include 465 youth and young adults (aged 6-30 years old) who sustain a TBI of any severity. An initial evaluative phase using the best available technology to evaluate eye and inner ear function will be performed, and compared with typical tests that are used in the clinic. If symptoms and functional problems remain 10 days after injury, participants will be randomly placed into a treatment group (including eye movement, inner ear-eye reflex and attention exercises as per our pilot studies) or a control group (typical rehabilitation). Success will be measured in terms of return to sport (mild TBI), achievement of goals (moderate and severe TBI) and quality of life. It is expected that this program will inform clinical practice and future research leading to a treatment program in TBI that includes multiple components.

ELIGIBILITY:
Inclusion Criteria:

* Mild TBI or moderate-severe TBI will be included

Exclusion Criteria:

-

Ages: 6 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
PedsQL | 8 weeks post intervention initiation
  Pediatric and adult Quality of Life
Head Thrust Test | 8 weeks post-intervention initiation
  Vestibulo-Ocular Reflex

CONTACTS AND LOCATIONS:
Locations (4):
- Canada (2):
  - Sport Injury Prevention Research Centre, Faculty of Kinesiology, University of Calgary,, Calgary, Alberta
  - Montreal Children's Hospital, MUHC, Montreal, Quebec
- Service de Rééducation des Pathologies Neurologiques de l'Enfant - Pôle de Rééducation et Réadaptation de l'Enfant Hôpitaux de Saint Maurice, Saint-Maurice, France
- Department of Physical Therapy, School of Health Professions, Sackler Faculty of Medicine, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sorek G, Shaklai S, Gagnon I, Schneider K, Chevignard M, Stern N, Fadida Y, Kalderon L, Katz-Leurer M. Impact of Subarachnoid Hemorrhage on the Cardiac Autonomic Function During Rehabilitation in Children After Severe Traumatic Brain Injury. Neurotrauma Rep. 2023 Jul 14;4(1):458-462. doi: 10.1089/neur.2023.0032. eCollection 2023. PMID 37475976
- [Derived] Sorek G, Gagnon I, Schneider K, Chevignard M, Stern N, Fadida Y, Kalderon L, Shaklai S, Katz-Leurer M. The Cardiac Autonomic Response Recovery to the Modified Tilt Test in Children Post Moderate-Severe Traumatic Brain Injury. Brain Inj. 2022 Jul 3;36(8):1033-1038. doi: 10.1080/02699052.2022.2110942. Epub 2022 Aug 15. PMID 35971307
- [Derived] Sorek G, Gagnon I, Schneider K, Chevignard M, Stern N, Fadida Y, Kalderon L, Shaklai S, Katz-Leurer M. The integrated functions of the cardiac autonomic and vestibular/oculomotor systems in adolescents following severe traumatic brain injury and typically developing controls. Brain Inj. 2020 Sep 18;34(11):1480-1488. doi: 10.1080/02699052.2020.1807055. Epub 2020 Aug 18. PMID 32809873